CLINICAL TRIAL: NCT02844790
Title: A Trial Investigating the Pharmacokinetic Properties of Insulin Degludec/Insulin Aspart in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN5401-1984; U1111-1173-7678 (Other: WHO)
Record Dates: First submitted 2016-07-22; First posted 2016-07-26 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Healthy
MeSH Terms: interventions — insulin degludec, insulin aspart drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IDegAsp (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart

INTERVENTIONS:
Drug: insulin degludec/insulin aspart — A single dose of IDegAsp will be administered subcutaneously (s.c., under the skin).

SUMMARY:
This trial is conducted in Asia. The aim of this trial is to investigate the pharmacokinetic (the exposure of the trial drug in the body) properties of insulin degludec/insulin aspart in healthy Chinese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Chinese subject aged 18-45 years (both inclusive)
* Considered generally healthy upon completion of medical history, physical examination, vital signs and electrocardiogram (ECG), as judged by the investigator
* Body mass index 19.0-24.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* A history of any illness that, in the opinion of the investigator, might confound the results of the trial or pose risk in administering the trial product to the subject
* Subject who has donated any blood or plasma in the past month or more than 400 mL within 3 months prior to screening
* Smoking more than 5 cigarettes (including nicotine substitute products), or the equivalent, per

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-07-26 (Actual); Primary Completion 2016-09-26 (Actual); Study Completion 2016-09-27 (Actual)

PRIMARY OUTCOMES:
Area under the serum insulin degludec concentration-time curve | From 0 to 120 hours after single dose
Area under the serum insulin aspart concentration-time curve | From 0 to 12 hours after single dose

SECONDARY OUTCOMES:
Maximum observed serum insulin degludec concentration | After single dose (within 0 to 120 hours after dosing)
Maximum observed serum insulin aspart concentration | After single dose (within 0 to 12 hours after dosing)
Time to maximum observed serum insulin degludec concentration | After single dose (within 0 to 120 hours after dosing)
Time to maximum observed serum insulin aspart concentration | After single dose (within 0 to 12 hours after dosing)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Beijing, China

REFERENCES:
- [Background] Aixin S, Yang L, Panpan X, Qi W , Lei Y, Hongfei X, Ran LZ, Haahr H. A study investigating the pharmacokinetic properties of insulin degludec/insulin aspart in healthy Chinese subjects. Diabetes Manag. 2019; 9 (2): 48-56.
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com